CLINICAL TRIAL: NCT00696423
Title: Immunogenicity and Reactogenicity Study of GlaxoSmithKline Biologicals' Infanrix™/Hib Vaccine Administered as a Booster Dose to 18-24 Months Old Children
Brief Title: Immunogenicity and Safety of GSK Biologicals' Infanrix/Hib in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111535
Record Dates: First submitted 2008-06-05; First posted 2008-06-12 (Estimated); Results first posted 2009-08-26 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2016-10

CONDITIONS: Acellular Pertussis; Diphtheria; Tetanus
Keywords: Infanrix/Hib; Chinese children
MeSH Terms: conditions — Diphtheria; Tetanus | interventions — Diphtheria-Tetanus-acellular Pertussis Vaccines; Hiberix

ARMS (2):
- Infanrix/Hib Single Injection Group (Experimental): Subjects received 1 dose of Infanrix™ extemporaneously mixed with Hiberix™.
  Interventions: Biological: Infanrix™; Biological: Hiberix™
- Infanrix + Hiberix Separate Injection Group (Active Comparator): Subjects received two separate injections, one of Infanrix™ and one of Hiberix™.
  Interventions: Biological: Infanrix™; Biological: Hiberix™

INTERVENTIONS:
Biological: Infanrix™ — Intramuscular injection, one dose
Biological: Hiberix™ — Intramuscular injection, one dose

SUMMARY:
This protocol posting deals with objectives & outcome measures of the booster phase. The objectives & outcome measures of the primary phase are presented in a separate protocol posting (NCT number = NCT00412854). This Phase IIIB study will compare GSK Biologicals' DTPa/Hib vaccine to separately administered DTPa and Hib vaccines in Chinese children 18 to 24 months of age, in terms of safety and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* Subjects should have completed the full three-dose primary vaccination course in study 104567.
* A male or female child between, and including, 18 and 24 months of age at the time of the booster vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding booster vaccination, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the booster dose.
* Administration of a vaccine not foreseen by the study protocol within 30 days prior to vaccination, or planned administration during the study period, with the exception of measles or combined measles, mumps and rubella (MMR) vaccination.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Previous booster vaccination against diphtheria, tetanus, pertussis and/or Haemophilus influenzae type b diseases since the end of the primary study.
* History of diphtheria, tetanus, pertussis and/or Haemophilus influenzae type b diseases.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s).
* Major congenital defects or serious chronic illness.
* History of any progressive neurological disorders or seizures.
* Acute disease and/or fever at time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the booster dose or planned administration during the study period.
* Occurrence of any of the following adverse events (AEs) after previous administration of a diphtheria-tetanus-pertussis (DTP) vaccine:

  * Hypersensitivity reaction due to any component of the vaccine.
  * Encephalopathy.
  * Fever ≥ 40.0 °C (axillary temperature) within 48 hours of vaccination.
  * Collapse or shock-like state within 48 hours of vaccination.
  * Persistent, inconsolable crying occurring within 48 hours of vaccination and lasting ≥ 3 hours.
  * Seizures with or without fever occurring within 3 days of vaccination.

Ages: 18 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 467 (Actual)
Dates: Start 2008-06-07; Primary Completion 2008-07-26 (Actual); Study Completion 2008-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- China (3):
  - GSK Investigational Site, Liucheng County, Guangxi
  - GSK Investigational Site, Mengshan
  - GSK Investigational Site, Wuzhou

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 111535 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111535 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111535 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111535 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111535 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111535 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111535 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Infanrix/Hib Single Injection Group: Subjects received 1 dose of Infanrix extemporaneously mixed with Hiberix.
- Infanrix + Hiberix Separate Injection Group: Subjects received two separate injections, one of Infanrix and one of Hiberix.
Period: Overall Study
Arm/Group | Infanrix/Hib Single Injection Group | Infanrix + Hiberix Separate Injection Group
Started | 244 | 223
Completed | 244 | 218
Not Completed | 0 | 5
Not completed — Lost to Follow-up | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infanrix/Hib Single Injection Group | Infanrix + Hiberix Separate Injection Group | Total
Number analyzed (Participants) | 244 | 223 | 467
Age, Continuous [Mean (Standard Deviation); unit: months] | 19.2 (0.79) | 19.2 (0.75) | 19.2 (0.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 111 | 224
  Male | 131 | 112 | 243

OUTCOME MEASURES:

1. Primary Outcome: Anti-polyribosyl-ribitol-phosphate (PRP) Antibody Concentrations
Description: Geometric mean concentrations are given in microgram per milliliter (μg/mL).
Time Frame: One month after booster vaccination
Population: Analysis was performed on the According To Protocol (ATP) cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Infanrix/Hib Single Injection Group | Infanrix + Hiberix Separate Injection Group
Number analyzed (Participants) | 238 | 216
μg/mL | 34.428 [29.452 to 40.244] | 132.075 [112.563 to 154.970]

2. Primary Outcome: Anti-diphtheria Toxoid Antibody Concentrations
Description: Geometric mean concentrations are given in international Unit per milliliter (IU/mL).
Time Frame: One month after booster vaccination
Population: Analysis was performed on the ATP cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Infanrix/Hib Single Injection Group | Infanrix + Hiberix Separate Injection Group
Number analyzed (Participants) | 237 | 214
IU/mL | 0.945 [0.905 to 0.987] | 0.926 [0.887 to 0.966]

3. Primary Outcome: Anti-tetanus Toxoid Antibody Concentrations
Description: Geometric mean concentrations are given in IU/mL.
Time Frame: One month after booster vaccination
Population: Analysis was performed on the ATP cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Infanrix/Hib Single Injection Group | Infanrix + Hiberix Separate Injection Group
Number analyzed (Participants) | 237 | 214
IU/mL | 7.455 [6.881 to 8.077] | 10.104 [9.080 to 11.242]

4. Primary Outcome: Anti-pertussis Toxoid (PT), Anti-filamentous Haemagglutinin (FHA) and Anti-pertactin (PRN) Antibody Concentrations
Description: Geometric mean concentrations are given in Enzyme-Linked Immuno Sorbent Assay (ELISA) unit per milliliter (EL.U/mL).
Time Frame: One month after booster vaccination
Population: Analysis was performed on the ATP cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Infanrix/Hib Single Injection Group | Infanrix + Hiberix Separate Injection Group
Number analyzed (Participants) | 239 | 216
EL.U/mL
  Anti-PT | 52.2 [48.1 to 56.7] | 55.8 [51.7 to 60.3]
  Anti-FHA | 93.3 [82.6 to 105.4] | 92.8 [83.3 to 103.4]
  Anti-PRN | 235.9 [208.7 to 266.5] | 241.6 [213.6 to 273.2]

5. Primary Outcome: The Number of Subjects Seroprotected for Anti-PRP, Anti-diphtheria and Anti-tetanus Antibodies and Seropositive for Anti-PT, Anti-FHA and Anti-PRN Antibodies
Description: Assay cut-offs indicating seroprotection or seropositivity for the different antigens were the following: anti-PRP antibody concentrations ≥ 0.15 µg/mL, anti-diphtheria and anti-tetanus antibody concentrations ≥ 0.1 IU/mL, anti-PT, anti-FHA and anti-PRN antibody concentrations ≥ 20 EL.U/mL.
Time Frame: One month after booster vaccination
Population: Analysis was performed on the ATP cohort for immunogenicity.
Measure: Number; unit: subjects
Arm/Group | Infanrix/Hib Single Injection Group | Infanrix + Hiberix Separate Injection Group
Number analyzed (Participants) | 239 | 216
subjects
  Seroprotection against PRP (n=238, 216) | 238 | 216
  Seroprotection against diphtheria (n=237, 214) | 237 | 214
  Seroprotection against tetanus (n=237, 214) | 237 | 214
  Seropositivity for anti-PT (n=239, 216) | 226 | 213
  Seropositivity for anti-FHA (n=239, 216) | 238 | 216
  Seropositivity for anti-PRN (n=239, 216) | 239 | 215

6. Secondary Outcome: Anti-PRP Antibody Concentrations
Description: Geometric mean concentrations are given in μg/mL.
Time Frame: Before booster vaccination
Population: Analysis was performed on the ATP cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Infanrix/Hib Single Injection Group | Infanrix + Hiberix Separate Injection Group
Number analyzed (Participants) | 237 | 216
μg/mL | 1.240 [1.085 to 1.418] | 2.461 [2.136 to 2.837]

7. Secondary Outcome: Anti-diphtheria Toxoid Antibody Concentrations
Description: Geometric mean concentrations are given in IU/mL.
Time Frame: Before booster vaccination
Population: Analysis was performed on the ATP cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Infanrix/Hib Single Injection Group | Infanrix + Hiberix Separate Injection Group
Number analyzed (Participants) | 237 | 214
IU/mL | 0.055 [0.053 to 0.058] | 0.054 [0.052 to 0.057]

8. Secondary Outcome: Anti-tetanus Toxoid Antibody Concentrations
Description: Geometric mean concentrations are given in IU/mL.
Time Frame: Before booster vaccination
Population: Analysis was performed on the ATP cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Infanrix/Hib Single Injection Group | Infanrix + Hiberix Separate Injection Group
Number analyzed (Participants) | 237 | 214
IU/mL | 0.219 [0.195 to 0.247] | 0.311 [0.274 to 0.353]

9. Secondary Outcome: Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations
Description: Geometric mean concentrations are given in EL.U/mL.
Time Frame: Before booster vaccination
Population: Analysis was performed on the ATP cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Infanrix/Hib Single Injection Group | Infanrix + Hiberix Separate Injection Group
Number analyzed (Participants) | 239 | 216
EL.U/mL
  Anti-PT | 10.0 [10.0 to 10.0] | 10.0 [10.0 to 10.1]
  Anti-FHA | 10.1 [10.0 to 10.2] | 10.3 [9.9 to 10.7]
  Anti-PRN | 10.2 [10.0 to 10.4] | 10.3 [10.0 to 10.5]

10. Secondary Outcome: The Number of Subjects Seroprotected for Anti-PRP, Anti-diphtheria and Anti-tetanus Antibodies and Seropositive for Anti-PT, Anti-FHA and Anti-PRN Antibodies
Description: as for outcome 5
Time Frame: Before booster vaccination
Population: Analysis was performed on the ATP cohort for immunogenicity.
Measure: Number; unit: subjects
Arm/Group | Infanrix/Hib Single Injection Group | Infanrix + Hiberix Separate Injection Group
Number analyzed (Participants) | 239 | 216
subjects
  Seroprotection against PRP (n= 237, 216) | 236 | 216
  Seroprotection against diphtheria (n= 237, 214) | 21 | 16
  Seroprotection against tetanus (n= 237, 214) | 209 | 198
  Seropositivity for anti-PT (n= 239, 216) | 0 | 1
  Seropositivity for anti-FHA (n= 239, 216) | 2 | 3
  Seropositivity for anti-PRN (n= 239, 216) | 3 | 4

11. Secondary Outcome: Number of Subjects Reporting Solicited Local and General Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling. Solicited general symptoms assessed include drowsiness, fever, irritability, and loss of appetite.
Time Frame: During the 4-day follow-up period after booster vaccination
Population: Analysis was performed on subjects from the Total Vaccinated Cohort with a documented dose.
Measure: Number; unit: subjects
Arm/Group | Infanrix/Hib Single Injection Group | Infanrix + Hiberix Separate Injection Group
Number analyzed (Participants) | 244 | 220
subjects
  Pain | 26 | 26
  Redness | 16 | 8
  Swelling | 9 | 1
  Drowsiness | 26 | 20
  Fever | 73 | 93
  Irritability | 43 | 46
  Loss of appetite | 40 | 39

12. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AE)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: During the 31-day follow-up period after booster vaccination
Measure: Number; unit: subjects
Arm/Group | Infanrix/Hib Single Injection Group | Infanrix + Hiberix Separate Injection Group
Number analyzed (Participants) | 244 | 223
subjects | 66 | 56

13. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAE)
Description: An SAE is any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in isability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: During the 31-day follow-up period after booster vaccination
Measure: Number; unit: subjects
Arm/Group | Infanrix/Hib Single Injection Group | Infanrix + Hiberix Separate Injection Group
Number analyzed (Participants) | 244 | 223
subjects | 1 | 3

ADVERSE EVENTS:
Arm/Group | Infanrix/Hib Single Injection Group | Infanrix + Hiberix Separate Injection Group
Serious Adverse Events (participants affected / at risk) | 1 | 3
Other Adverse Events (participants affected / at risk) | 133/244 | 127/223
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Infanrix/Hib Single Injection Group | Infanrix + Hiberix Separate Injection Group
Bronchopneumonia (Infections and infestations) | 1/240 | 2/223
Bronchitis (Infections and infestations) | 0/240 | 1/223
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Infanrix/Hib Single Injection Group (N=244) | Infanrix + Hiberix Separate Injection Group (N=223)
Pain at injection site (General disorders) | 26 | 26
Redness at injection site (General disorders) | 16 | 8
Drowsiness (General disorders) | 26 | 20
Fever (General disorders) | 73 | 93
Irritability (General disorders) | 43 | 46
Loss of appetite (General disorders) | 40 | 39
Nasopharyngitis (Infections and infestations) | 39 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.